CLINICAL TRIAL: NCT00139854
Title: A Multicenter, Open-Label, Randomized Crossover Trial to Assess Subject Preference for Alprazolam Orally Disintegrating Tablets Compared to Conventional Alprazolam Tablets in Subjects With Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SP829
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2009-09

CONDITIONS: ANXIETY
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Drug: Alprazolam orally disintegrating tablets

SUMMARY:
This was a multicenter, open-label, randomized crossover trial comparing two treatments, Alprazolam ODT versus conventional alprazolam tablets, in subjects who were already taking conventional immediate-release alprazolam tablets for anxiety. The trial included five study visits (four periods of 7 3 -day duration): Screening (Visit 1), Treatment Period 1 (Visit 2), Treatment Period 2 (Visit 3), Final Visit (Visit 4), and Follow-up (Visit 5 [telephone visit]). At Visit 1, following screening, eligible subjects continued to take their own conventional alprazolam as prescribed by their physician. At Visit 2, eligible subjects were randomized in approximately equal numbers to one of two treatment sequences: Alprazolam ODT/ conventional alprazolam or conventional alprazolam/ Alprazolam ODT. Subjects continued taking alprazolam in accordance with the treatment sequence to which they were assigned, at the same dose regimen as their own prescribed alprazolam. At Visit 3, subjects crossed over to the alternate treatment until Visit 4. At Visit 4, subjects completed the Subject Preference Questionnaire, and a physical examination and clinical laboratory tests were performed. At the end of Visit 4, subjects resumed taking their own conventional alprazolam. The site made a follow-up telephone call 7 - 3 days after Visit 4 to assess the subject's health status.

DETAILED DESCRIPTION:
See approved Package Insert for Adverse Event information.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with conventional alprazolam

Exclusion Criteria:

* Dose of greater than 10 mg

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States